CLINICAL TRIAL: NCT06326307
Title: Effectiveness of Puppet Modeling Technique on Children Undergoing Stressful Dental Procedures' Randomized Clinical Crossover Trial
Brief Title: Effectiveness of Puppet Modeling Technique on Children Undergoing Stressful Dental Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Layla Khogeer, Dr, King Abdulaziz University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 247-05-21
Record Dates: First submitted 2024-03-05; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Behavioral Guidance in Pediatric Dentistry
Keywords: behavioral guidance; Pediatric dentistry; puppet; tell show and do

STUDY DESIGN:
Intervention Model Description: * Group I : Children who received puppet behavior guidance during their first visit and tell-show-do guidance in their second visit, 2 weeks later. (P-TSD)
  * Group II: Children who received the tell-show-do behavior guidance during their first visit and puppet behavioral guidance in their second visit, 2 weeks later.(TSD-P)
Who Masked: Outcomes Assessor
Masking Description: Two evaluators, who are blinded to the experimented techniques, watched recorded videos of both groups separately and gave their behavior assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Children who received puppet behavior guidance during their first visit and tell-show-do guidance in their second visit, 2 weeks later. (P-TSD)
  Interventions: Behavioral: Tell Show and Do Guidance; Behavioral: Puppet Guidance
- Group 2 (Experimental): Children who received the tell-show-do behavior guidance during their first visit and puppet behavioral guidance in their second visit, 2 weeks later.(TSD-P)
  Interventions: Behavioral: Tell Show and Do Guidance; Behavioral: Puppet Guidance

INTERVENTIONS:
Behavioral: Tell Show and Do Guidance — In this technique, the dentist tells explains the procedure using the Tell show and do method.
Behavioral: Puppet Guidance — In this technique, the dentist using the puppet to explains the procedure.

SUMMARY:
The goal of this RCT is to compare puppet modeling technique vs tell show and do on children undergoing stressful dental procedures'

* The main question[s] it aims to answer are:

  1. To compare the effect of puppet modeling vs tell show and do on the cooperation of children during the administration of local anesthesia.
  2. To compare the effect of puppet modeling vs tell show and do on the anxiety level of children during the administration of local anesthesia.

type of study: clinical trial participant population/health conditions: Healthy

In this randomized crossover clinical trial, study subjects were randomly allocated into two groups:

* Group I : Children who received puppet behavior guidance during their first visit and tell-show-do guidance in their second visit, 2 weeks later. (P-TSD)
* Group II : Children who received the tell-show-do behavior guidance during their first visit and puppet behavioral guidance in their second visit, 2 weeks later.(TSD-P)

DETAILED DESCRIPTION:
Aim of the Study: The aim of this research is to compare the effectiveness of tell show and do (TSD) vs puppet play therapy on children's behavior during the administration of local anesthesia.

Materials and Methods: This was a randomized crossover clinical trail that was conducted at King Abdulaziz University Faculty of Dentistry for a period of 12 months starting from Jan 2023 to Dec 2023 on 41 children (aged 3-7 years) randomly divided into two groups of. Group I (23 children): Children who received the TSD behavior guidance during their first visit and puppet play therapy in their second visit 2 weeks later. Group II (18 children): Children who received puppet play therapy during their first visit and TSD guidance in their second visit 2 weeks later. The anxiety level was determined using Facial Index Scale(FIS) and Venham anxiety rating scale and pulse rate (PR) at the beginning, middle and the end of each anesthesia administration. Patient behavior was also scored using Frankl behavior rating scale (FBRS) , Venham behavior rating scale. The FLACC scale was used to assess pain.

ELIGIBILITY:
Inclusion Criteria:

* • Children having no previous experience of local anesthesia

  * Children aged 3-8 years old
  * Children with negative history of any particular underlying disease.

Exclusion Criteria:

* • Children who needed procedures with no local anesthesia.

  * Children who were allergic to local anesthesia.
  * Children who were indicated for advanced behavioral guidance.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Heart rate | through study completion, an average of 1 year
  The heart rate was measured throughout the procedure using Gibson finger oximeter. Three readings were recorded. One before the administration of local anesthesia, one during the injection and one immediately after.
Facial Image Scale | through study completion, an average of 1 year
  The FIS comprises a row of five faces ranging from (1) very happy to (5) very unhappy. It is simple, efficient measure of anxiety in very young children than other measures of anxiety that depend on the cognitive ability of the child
Vehnam Anxiety Rating Scale | through study completion, an average of 1 year
  The Vehnam Anxiety Rating Scale was used in this clinical trial to measure the patient's situational dental anxiety. This scale is an interval rating scale with the interval ranging from 0 (the least anxious score) to 5 (the most anxious
Frankl behavior rating scale | through study completion, an average of 1 year
  It classifies child behavior into four groups according to the child's attitude during dental treatment: (4)Definitely positive, (3) Positive, (2) Negative, and (1) Definitely negative.
FLACC Pain scale | through study completion, an average of 1 year
  Pain is assessed through observation of 5 categories including face, legs, activity, cry, and consolability. Each category will be given a score ranging from 0 to 2. The final score is calculated by adding up the scores of the five categories for a final score out of 10.
Venham Scale of Dental behavior | through study completion, an average of 1 year
  The Venham Scale of Dental behavior is an interval rating scale with the interval ranking from 0 (extremely cooperative) to 5 (extremely uncooperative).

CONTACTS AND LOCATIONS:
Locations (1):
- King Abulaziz university dental hospital, Jeddah, Mecca Region, Saudi Arabia

REFERENCES:
- [Derived] Khogeer LN, Sabbagh HJ, Felemban OM, Farsi NM. Puppet play therapy in emergency pediatric dental clinic. A randomized clinical trial. BMC Pediatr. 2025 Jul 2;25(1):503. doi: 10.1186/s12887-025-05849-5. PMID 40604606